CLINICAL TRIAL: NCT01263067
Title: Lifespan Integration Therapy for Posttraumatic Stress Disorder of Adults Involved in an Auto Accident
Brief Title: Lifespan Integration for Posttraumatic Stress Disorder From an Auto Accident
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Argosy University (Other)
Responsible Party: Principal Investigator, Elana Rosencrantz, Student, Argosy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-10
Record Dates: First submitted 2010-12-15; First posted 2010-12-20 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; PTSD; Car Accident; Auto Accident; Lifespan Integration
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifespan Integration Therapy (LI) (Experimental)
  Interventions: Behavioral: Lifespan Integration Therapy
- Waitlist Control- Lifespan Integration (Active Comparator)
  Interventions: Behavioral: Lifespan Integration- Control

INTERVENTIONS:
Behavioral: Lifespan Integration Therapy — LI treatment guides the client to imaginally visit past memories, and then leads her or him forward through time to the present using a concept referred to as the time line. Beginning with the individual's memories from the traumatic experience, the time line first follows memories from the days and weeks after the trauma, then season by season to the present, and is reviewed in ongoing sessions as increasing details of the traumatic event are uncovered.
  Arms: Lifespan Integration Therapy (LI)
Behavioral: Lifespan Integration- Control — Participants selected for the control group will be treated 4 weeks following initial contact. Treatment is the same as for the Experimental Group.
  Arms: Waitlist Control- Lifespan Integration

SUMMARY:
The purpose of this study is to evaluate if lifespan integration (LI) therapy reduces posttraumatic stress symptoms following a motor vehicle accident (MVA) trauma

DETAILED DESCRIPTION:
Studies estimate a substantial proportion of MVA survivors, ranging from 9.4% to 59.9%, will develop PTSD following an accident (Blanchard & Hickling, 2004). Based on conservative estimates, past research, indicates that MVA-related PTSD may affect 2.5 to 7 million persons in the United States (Blanchard & Hickling). Furthermore, two seminal epidemiological studies (Kessler et al., 1995; Norris, 1992) that focused on causes of adult PTSD identified MVAs as the most frequent trauma resulting in PTSD. For these reasons, MVA-resultant PTSD represents a significant public health problem that needs not only to be thoroughly understood, but addressed with successful mental health treatment options (Beck & Coffey, 2007; Blanchard & Hickling, 1997, 2004; Bryant et al., 1998; Taylor et al., 1999; Taylor et al., 2001). Although there is empirical literature on the treatment of PTSD following an MVA, additional efficacious and rigorously conducted studies with statistical underpinnings are required to determine the results that can be expected from alternative models of care (Beck & Coffey; Blanchard & Hickling, 1997, 2004).

ELIGIBILITY:
Inclusion Criteria:

* Involved in or witnessed a car accident at least 6 months ago.
* PTSD or distress or impairment in important areas of functioning following the car accident

Exclusion Criteria:

* moderate or severe head injury
* current mental health treatment for the MVA-related problem
* severe chronic pre-injury mental health problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Clinicians Administered PTSD Scale | following the final treatment session (average of 6 weeks from treatment start date)
  Participants will be assessed with the CAPS following the final treatment session (up to 5 treatment sessions).

SECONDARY OUTCOMES:
Personality Assessment Inventory | following the final treatment session (average of 6 weeks from treatment start date)

CONTACTS AND LOCATIONS:
Overall Officials: Frances Parks, PhD, Study Chair — Argosy University Seattle
Locations (1):
- Argosy University Seattle, Seattle, Washington, United States

REFERENCES:
- [Background] Pace, P. (2007). Lifespan integration: Connecting ego states through time (fourth ed.). Roslyn, WA: Peggy Pace.
- See also: Related Info — http://www.lifespanintegration.com